CLINICAL TRIAL: NCT03332095
Title: Phase I/II Study of the Pharmacokinetics, Safety and Tolerability of Doravirine (MK-1439) and Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (MK-1439A) in HIV-1-Infected Children and Adolescents
Brief Title: Evaluating the Pharmacokinetics, Safety, and Tolerability of Doravirine (MK-1439) and Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (MK-1439A) in HIV-1-Infected Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2014; 34150 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — doravirine; Anti-Retroviral Agents; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: DOR (Experimental): Participants received a single dose of DOR at study entry (Day 0).
  Interventions: Drug: Doravirine (DOR); Drug: Antiretroviral (ARV) medications
- Cohort 2: DOR/3TC/TDF (Experimental): Participants received DOR/3TC/TDF from Day 0 through Week 96.
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF)

INTERVENTIONS:
Drug: Doravirine (DOR) — 100 mg of DOR administered orally
  Other Names: MK-1439
  Arms: Cohort 1: DOR
Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) — DOR/3TC/TDF administered orally as a fixed-dose combination (as a tablet, 100 mg/300 mg/300 mg) once daily
  Other Names: MK-1439A
  Arms: Cohort 2: DOR/3TC/TDF
Drug: Antiretroviral (ARV) medications — Participants in Cohort 1 received a combination of dolutegravir (DTG) or raltegravir (RAL) plus two nucleoside reverse transcriptase inhibitors (NRTIs). The ARV drugs were prescribed by participants' own health care providers and were not provided by the study.
  Other Names: ARVs
  Arms: Cohort 1: DOR

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics, safety, and tolerability of doravirine (also called MK-1439 or DOR) and doravirine/lamivudine/tenofovir disoproxil fumarate (also called MK-1439A or DOR/3TC/TDF) in HIV-1-infected children and adolescents.

DETAILED DESCRIPTION:
This study evaluated the pharmacokinetics (PK), safety, and tolerability of DOR and DOR/3TC/TDF in HIV-1-infected children and adolescents.

This study was conducted in two cohorts: Cohort 1 and Cohort 2. At study entry (Day 0), participants in Cohort 1 received a single dose of DOR added to their current HIV regimens. (The antiretroviral drugs in their current HIV regimens were not be provided by the study.) Participants in Cohort 1 underwent intensive PK evaluations, and had an additional study visit at Week 2.

The study team in consultation with a Study Monitoring Committee evaluated data from Cohort 1 before enrolling participants in Cohort 2. Participants in Cohort 2 received DOR/3TC/TDF once daily from Day 0 through Week 96. They had study visits at Weeks 1, 2, 4, 8, 12, 16, 24, 36, 48, 64, 80, and 96. Study visits included physical examinations, PK evaluations, and blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than or equal 35 kg at entry
* If not of legal age to provide independent informed consent: Parent or guardian was willing and able to provide written informed consent for study participation; in addition, when applicable per local Institutional Review Board / Ethics Committee (IRB/EC) policies and procedures, potential participant was willing and able to provide written informed assent for study participation. If of legal age to provide independent informed consent as determined by site Standard Operating Procedures (SOPs) and consistent with site IRB/EC policies and procedures: Potential participant was willing and able to provide written informed consent for study participation
* Confirmed HIV-1-infection based on documented testing of two samples collected at different time points. More information on this criterion can be found in the protocol.
* Antiretroviral therapy (ART) exposure, virologic suppression, and resistance requirements, as follows:

Cohort 1

* ART exposure requirements, based on individual or parent/guardian's report and, if available, confirmed by medical records:
* At entry, receiving combination ART with raltegravir (RAL) or dolutegravir (DTG) plus 2 nucleoside reverse transcriptase inhibitors (NRTIs); AND
* At entry, had not received non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitor (PIs), or cobicistat within the previous 30 days; AND
* Virologic suppression, as documented in medical records and as defined by:
* One or more HIV RNA polymerase chain reaction (PCR) result below the level of quantification (BLLQ) within 15 months prior to enrollment, AND
* If any HIV RNA PCR tests had been done within 3 months prior to enrollment, all results were below the level of quantification, AND
* HIV RNA PCR result less than 40 copies/mL at screening, performed as per the protocol.

Cohort 2 ART-naive

* ART exposure requirements, based on individual or parent/guardian's report and, if available, confirmed by medical records:
* At entry, received no antiretrovirals (ARVs) for treatment of HIV infection including investigational agents (prior receipt of ARVs for prevention of perinatal transmission was permitted); AND
* Screening genotypic resistance test results indicated susceptibility to doravirine (DOR), tenofovir disoproxil fumarate (TDF), and lamivudine (3TC) (see the protocol for more information; result must be available prior to enrollment), performed as per the protocol; AND
* If available, as documented in medical records, any prior genotypic resistance test result indicated susceptibility to DOR, TDF, and 3TC (see the protocol for more information).

Note: For individuals that were re-screened, the genotypic resistance test did not need to be repeated.

Cohort 2 ART-experienced

* ART exposure requirements, based on individual or parent/guardian's report and, if available, confirmed by medical records:
* No previous history of change in ARVs due to clinical or virologic failure, in the opinion of the site investigator or designee; AND
* Virologic suppression, as documented in medical record and as defined by:
* One or more HIV RNA PCR result BLLQ within 15 months prior to enrollment, AND
* If any HIV RNA PCR tests had been done within 3 months prior to enrollment, all results were below the level of quantification, AND
* HIV RNA PCR result less than 40 copies/mL at screening (see the protocol for more information); AND
* If available, as documented in medical records, any prior genotypic resistance test result indicated susceptibility to DOR, TDF, and 3TC (see the protocol for more information).

Note: This group of ARV-experienced, virologically suppressed participants were only enrolled once there was data from the adult switch studies indicating virologic efficacy and safety (see the protocol for more information). Sites were informed via a Clarification Memorandum when ART-experienced participants could be enrolled. A single, unconfirmed HIV-1 RNA result greater than or equal to the level of quantification but less than 500 copies/mL, between 3 and 15 months, prior to enrollment was not exclusionary as long as the other criteria for documentation of virologic suppression were met.

* Grade 2 or lower hemoglobin, aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase, and lipase on specimens obtained at screening
* For Cohort 2 only, grade 2 or lower creatinine, proteinuria, and glycosuria on specimens obtained at screening
* Estimated glomerular filtration rate (eGFR) greater than or equal to 60 mL/min/1.73 m^2, on specimens obtained at screening, based on the Schwartz equation. More information on this criterion can be found in the protocol.
* For females who had reached menarche or who were engaging in sexual activity (self-reported), negative pregnancy test at entry
* For females engaging in sexual activity that could lead to pregnancy (self-reported), agreed to use two effective, medically accepted birth control methods while on study and for two weeks after permanently discontinuing study drug
* For males engaging in sexual activity that could lead to pregnancy (self-reported), agreed to use condoms while on study and for two weeks after permanently discontinuing study drug
* Able and willing to swallow available formulation(s) (tablet or, as available, oral granules).

Exclusion Criteria:

• Evidence of decompensated liver disease manifested by the presence of or a history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy, or other signs or symptoms of advanced liver diseases.

Note: Individuals with chronic hepatitis B who had grade 2 or lower ALT and AST and had no significant impairment of hepatic synthetic function (significant impairment of hepatic synthetic function was defined as a serum albumin less than 2.8 mg/dL or an international normalized ratio (INR) greater than 1.7 in the absence of another explanation for the abnormal laboratory value) were eligible.

• For Cohort 2 only, detectable hepatitis C virus (HCV) by RNA PCR or current or planned treatment with direct antiviral agent for HCV.

Note: HCV antibody positivity but undetectable by HCV RNA PCR results were permitted.

* Presence of any active AIDS-defining opportunistic infection
* History of malignancy (ever), with the exception of localized malignancies such as squamous cell or basal cell carcinoma of the skin
* Clinical evidence of pancreatitis, as determined by the clinician (at entry)
* Use of nafcillin, dicloxacillin, or any of the prohibited medications, within 30 days prior to study entry (see the protocol for a complete list of prohibited medications)
* For females, currently breastfeeding an infant at entry
* Enrolled in another clinical trial of an investigational agent, device, or vaccine
* Unlikely to adhere to the study procedures or keep appointments, in the opinion of the site investigator or designee
* Used, or anticipates using, chronic systemic immunosuppressive agents or systemic interferon (e.g., for treatment of HCV infection) within 30 days prior to study entry.

Note: Systemic corticosteroids (e.g., prednisone or equivalent up to 2 mg/kg/day) for replacement therapy or short courses (less than or equal to 30 days) were permitted. See the protocol for a complete list of prohibited medications.

* Diagnosed with current active tuberculosis and/or was currently being treated with a rifampicin-containing regimen
* Individual had any other condition, that in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Melvin, MD, MPH, Study Chair — University of Washington, Seattle Children's Research Institute
Locations (8):
- United States (4):
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Soweto IMPAACT CRS, Johannesburg, Gauteng, South Africa
- Thailand (3):
  - Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai

REFERENCES:
- See also: Link to the IMPAACT 2014 study web page — http://impaactnetwork.org/studies/IMPAACT2014
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from July 2018 to February 2020. Participants were recruited from 8 medical clinics in the United States, Thailand and South Africa.
Pre-assignment Details: There was no randomization. Enrollment started with Cohort 1, then Cohort 2 was open.
Period: Overall Study
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Started | 10 | 45
Received at Least One Dose of Study Treatment | 9 | 45
Completed | 9 | 44
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study treatment.
Groups:
- Cohort 1: DOR: Participants received a single dose of DOR at study entry (Day 0).
  Doravirine (DOR): 100 mg of DOR administered orally
  Antiretroviral (ARV) medications: Participants in Cohort 1 received a combination of dolutegravir (DTG) or raltegravir (RAL) plus two nucleoside reverse transcriptase inhibitors (NRTIs). The ARV drugs were prescribed by participants' own health care providers and were not be provided by the study.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF | Total
Number analyzed (Participants) | 9 | 45 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.6) | 15.0 (1.6) | 14.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 26 | 28
  Male | 7 | 19 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 44 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 35 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 55.9 (15.8) | 53.8 (8.0) | 54.1 (9.5)
Weight Band (kg) [Count of Participants; unit: Participants]
  35 - <45 kg | 1 | 0 | 1
  ≥ 45 kg | 8 | 45 | 53
Region [Count of Participants; unit: Participants]
  Africa | 0 | 9 | 9
  Asia/Pacific | 0 | 35 | 35
  North America | 9 | 1 | 10
Class of Prior ARTs [Count of Participants; unit: Participants] — Various classes (types) of antiretroviral therapies (ART) that participants received prior to study entry.
  Participants
    Nucleoside Reverse Transcriptase Inhibitors (NRTI) | 9 | 43 | 52
    Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI) | 0 | 32 | 32
    Integrase Strand Transfer Inhibitors (INSTI) | 9 | 1 | 10
    Protease Inhibitors (PI) | 0 | 10 | 10
    Not Applicable | 0 | 2 | 2
Baseline Plasma HIV-1 RNA (copies/mL) [Count of Participants; unit: Participants]
  0 - <40 | 9 | 43 | 52
  40 - <500,000 | 0 | 0 | 0
  500,000 - <1,000,000 | 0 | 2 | 2
Duration of Prior ARTs [Mean (Standard Deviation); unit: days] | 614.2 (511.3) | 1882.3 (1649.6) | 1662.8 (1589.4)
CD4 Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 788.2 (203.9) | 717.8 (283.1) | 729.7 (270.9)
CD4% [Mean (Standard Deviation); unit: percent] | 36.2 (5.4) | 33.1 (9.1) | 33.6 (8.6)
HIV-1 log10 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 1.6 (0.0) | 1.8 (0.9) | 1.7 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Single-dose Area-under-the-curve (AUC0-∞) of Doravirine (DOR) (Cohort 1)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (WinNonlin version 6.3, Pharsight Corp., Mountain View, CA). Area under the curve (AUC) was determined using non-compartmental analyses and estimated by the linear up/log down trapezoidal rule, from time zero to infinity. Steady state AUC0-24 is equivalent to single dose AUC0-∞.
Time Frame: Measured during the entry (day 0) visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12, 24, 48 and 72 hours post-dose.
Population: Cohort 1 participants who received the study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 0
µM*hr | 34.8 (43.2) |

2. Primary Outcome: PK Parameter: Single-dose Maximum Concentration (Cmax) of DOR (Cohort 1)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (WinNonlin, version 6.3, Pharsight Corp., Mountain View, CA).
Time Frame: as for outcome 1
Population: Cohort 1 participants who received the study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 0
µM | 2.14 (25.9) |

3. Primary Outcome: PK Parameter: Single-dose 24 Hour-concentration (C24hr) of DOR (Cohort 1)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Cohort 1 participants who received the study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 0
nM | 514 (56.5) |

4. Primary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs) Assessed as Related to Study Drug
Description: Percentage and Clopper-Pearson 95% Confidence Interval (CI) of participants with Grade 3 or higher AEs judged by the medical clinic as related to the study drug. AEs were graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017 (see References).
Time Frame: Cohort 1: Measured from Day 0 through Week 2; Cohort 2: Measured from Day 0 through Week 24.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 45
percentage of participants | 0 [0 to 33.6] | 0 [0 to 7.9]

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Assessed as Related to Study Drug
Description: Percentage and Clopper-Pearson 95% CI of participants with SAEs judged by the medical clinic as related to the study drug. SAEs were reported according to Version 2.0 of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual) (see references).
Time Frame: Cohort 1: Measured from Day 0 through Week 2; Cohort 2: Measured from Day 0 through Week 24.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 45
percentage of participants | 0 [0 to 33.6] | 0 [0 to 7.9]

6. Primary Outcome: Percentage of Participants With Permanent Discontinuation of Study Drug Due to Adverse Events Assessed as Related to Study Drug
Description: Percentage and Clopper-Pearson 95% CI of participants with permanent discontinuation of study drug due to AEs judged by the medical clinic as related to the study drug.
Time Frame: Cohort 1: Measured from Day 0 through Week 2; Cohort 2: Measured from Day 0 through Week 24.
Population: Study Participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 45
percentage of participants | 0 [0 to 33.6] | 0 [0 to 7.9]

7. Primary Outcome: Percentage of Participants With Grade 5 Adverse Events (Death) Regardless of Relationship to Study Drug
Description: Percentage and Clopper-Pearson 95% CI of participants with Grade 5 AEs (death) regardless of relationship to study drug.
Time Frame: Cohort 1: Measured from Day 0 through Week 2; Cohort 2: Measured from Day 0 through Week 24.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 9 | 45
percentage of participants | 0 [0 to 33.6] | 0 [0 to 7.9]

8. Secondary Outcome: PK Parameter: AUC0-24hr of DOR (Cohort 2)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (WinNonlin, version 6.3, Pharsight Corp., Mountain View, CA). Area under the curve (AUC) was determined using non-compartmental analyses and estimated by the linear up/log down trapezoidal rule, from time zero to 24 hours. Intensive PK samples were collected for the first ten participants enrolled in Cohort 2.
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 2, 4, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
µM*hr |  | 22.9 (47.0)

9. Secondary Outcome: PK Parameter: AUC0-24hr of 3TC (Cohort 2)
Description: as for outcome 8
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
h.ng/mL |  | 11300 (27.9)

10. Secondary Outcome: PK Parameter: AUC0-24hr of Tenofovir (Cohort 2)
Description: as for outcome 8
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h.ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
h.ng/mL |  | 2550 (14.3)

11. Secondary Outcome: PK Parameter: Cmax of DOR (Cohort 2)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (WinNonlin, version 6.3, Pharsight Corp., Mountain View, CA). Cmax was projected from individual plasma concentration-time profiles using the non-parametric superposition function in WinNonLin v6.3. Intensive PK samples were collected for the first ten participants enrolled in Cohort 2.
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 2, 4, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
µM |  | 2.13 (42.7)

12. Secondary Outcome: PK Parameter: Cmax of 3TC (Cohort 2)
Description: as for outcome 11
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
ng/mL |  | 2100 (23.6)

13. Secondary Outcome: PK Parameter: Cmax of Tenofovir (Cohort 2)
Description: as for outcome 11
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
ng/mL |  | 293 (36.6)

14. Secondary Outcome: PK Parameter: C24hr of DOR (Cohort 2)
Description: Pharmacokinetic parameters were determined from plasma concentration-time profiles using non-compartmental methods (WinNonlin, version 6.3, Pharsight Corp., Mountain View, CA). C24hr was projected from individual plasma concentration-time profiles using the non-parametric superposition function in WinNonLin v6.3. Intensive PK samples were collected for the first ten participants enrolled in Cohort 2.
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 2, 4, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
nM |  | 282 (73.8)

15. Secondary Outcome: PK Parameter: C24hr of 3TC (Cohort 2)
Description: as for outcome 14
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
ng/mL |  | 66.3 (54.7)

16. Secondary Outcome: PK Parameter: C24hr of Tenofovir (Cohort 2)
Description: as for outcome 14
Time Frame: Measured at Week 1 visit. Blood samples were drawn at pre-dose, and at 1, 2, 4, 8, 12 and 24 hours post-dose.
Population: The first 10 participants enrolled in Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 10
ng/mL |  | 50.2 (9.4)

17. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 200 Copies/mL at Week 24 (Cohort 2)
Description: Virologic responses were assessed at week 24 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >200 copies/mL; otherwise participants with missing values were excluded.
Time Frame: Measured at week 24.
Population: Cohort 2 participants who received at least one dose of study treatment. Participants who discontinued study for reasons other than virologic failure were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 44
Percentage of participants |  | 97.7 [88.0 to 99.9]

18. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 200 Copies/mL at Week 48 (Cohort 2)
Description: Virologic responses were assessed at week 48 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >200 copies/mL; otherwise participants with missing values were excluded.
Time Frame: Measured at week 48.
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 44
Percentage of participants |  | 97.7 [88.0 to 99.9]

19. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 200 Copies/mL at Week 96 (Cohort 2)
Description: Virologic responses were assessed at week 96 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >200 copies/mL; otherwise participants with missing values were excluded.
Time Frame: Measured at week 96.
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 42
Percentage of participants |  | 92.9 [80.5 to 98.5]

20. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 50 Copies/mL at Week 24 (Cohort 2)
Description: Virologic responses were assessed at week 24 as percentage of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >50 copies/mL. Otherwise participants with missing values were excluded.
Time Frame: Measured at week 24.
Population: Cohort 2 participants who received at least one dose of study treatment. Participants who discontinued study for reasons other than virologic failure were excluded. One participant whose sample was diluted due to low volume, resulting in increased assay limit of quantification from 40 to 200 copies/mL was excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
Percentage of participants |  | 97.7 [87.7 to 99.9]

21. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 50 Copies/mL at Week 48 (Cohort 2)
Description: Virologic responses were assessed at week 48 as percentage of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >50 copies/mL. Otherwise participants with missing values were excluded.
Time Frame: Measured at week 48.
Population: Cohort 2 participants who received at least one dose of study treatment. Participants who discontinued study for reasons other than virologic failure were excluded. Two participants whose sample was diluted due to low volume, resulting in increased assay limit of quantification from 40 to 200 copies/mL were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 42
Percentage of participants |  | 97.6 [87.4 to 99.9]

22. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 50 Copies/mL at Week 96 (Cohort 2)
Description: Virologic responses were assessed at week 96 as percentage of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >50 copies/mL. Otherwise participants with missing values were excluded.
Time Frame: Measured at week 96.
Population: Cohort 2 participants who received at least one dose of study treatment. Participants who discontinued study for reasons other than virologic failure were excluded. Two participant whose sample was diluted due to low volume, resulting in increased assay limit of quantification from 40 to 200 copies/mL were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 40
Percentage of participants |  | 92.5 [79.6 to 98.4]

23. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 40 Copies/mL at Week 24 (Cohort 2)
Description: Virologic responses were assessed at week 24 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >40 copies/mL; Otherwise participants with missing values were excluded.
Time Frame: Measured at week 24.
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
Percentage of participants |  | 97.7 [87.7 to 99.9]

24. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 40 Copies/mL at Week 48 (Cohort 2)
Description: Virologic responses were assessed at week 48 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >40 copies/mL; Otherwise participants with missing values were excluded.
Time Frame: Measured at week 48.
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 42
Percentage of participants |  | 97.6 [87.4 to 99.9]

25. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than 40 Copies/mL at Week 96 (Cohort 2)
Description: Virologic responses were assessed at week 96 as percentage (%) of participants and Clopper-Pearson 95% CI. Missing values were considered as failures for participants with missing data due to discontinuation of study drug as a result of virologic failure or for non-treatment related reasons with last available RNA >40 copies/mL; Otherwise participants with missing values were excluded.
Time Frame: Measured at week 96.
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 40
Percentage of participants |  | 92.5 [79.6 to 98.4]

26. Secondary Outcome: Summary of log10 Drop From Baseline to Week 24 in Plasma HIV-1 RNA (ART-naive Participants) (Cohort 2)
Description: The differences between log10 HIV RNA at Week 24 minus at Day 0 are summarized.
Time Frame: Measured at Day 0 and week 24.
Population: Cohort 2 participants who were ART-naive.
Measure: Mean (95% Confidence Interval); unit: Log10 plasma HIV-1 RNA
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 2
Log10 plasma HIV-1 RNA |  | -2.6 [-5.8 to 19.0]

27. Secondary Outcome: Summary of log10 Drop From Baseline to Week 48 in Plasma HIV-1 RNA (ART-naive Participants) (Cohort 2)
Description: The differences between log10 HIV RNA at Week 48 minus at Day 0 are summarized.
Time Frame: Measured at Day 0 and week 48.
Population: Cohort 2 participants who were ART-naive.
Measure: Mean (95% Confidence Interval); unit: Log10 plasma HIV-1 RNA
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 2
Log10 plasma HIV-1 RNA |  | -2.1 [-5.8 to 26.1]

28. Secondary Outcome: Summary of log10 Drop From Baseline to Week 96 in Plasma HIV-1 RNA (ART-naive Participants) (Cohort 2)
Description: The differences between log10 HIV RNA at Week 96 minus at Day 0 are summarized.
Time Frame: Measured at Day 0 and week 96.
Population: Cohort 2 participants who were ART-naive.
Measure: Mean (95% Confidence Interval); unit: Log10 plasma HIV-1 RNA
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 1
Log10 plasma HIV-1 RNA |  | -4.3

29. Secondary Outcome: Summary of Changes in CD4 Count From Baseline to Week 24 (Cohort 2)
Description: The mean difference is calculated as CD4 count at Week 24 minus CD4 count at Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 24.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 24 timepoints.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
cells/mm^3 |  | 84.8 [21.1 to 148.4]

30. Secondary Outcome: Summary of Changes in CD4 Count From Baseline to Week 48 (Cohort 2)
Description: The mean differences is calculated as CD4 count at Week 48 minus CD4 count at Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 48.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 48 timepoints.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
cells/mm^3 |  | 80.1 [14.2 to 146.0]

31. Secondary Outcome: Summary of Changes in CD4 Count From Baseline to Week 96 (Cohort 2)
Description: The mean difference is calculated as CD4 count at Week 96 minus CD4 count at Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 96.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 96 timepoints.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 38
cells/mm^3 |  | 42.5 [-31.1 to 116.1]

32. Secondary Outcome: Summary of Changes in CD4% From Baseline to Week 24 (Cohort 2)
Description: The mean difference is calculated as CD4% at Week 24 minus CD4% at Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 24.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 24 timepoints.
Measure: Mean (95% Confidence Interval); unit: Percent of total lymphocytes
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
Percent of total lymphocytes |  | -1.5 [-2.8 to -0.2]

33. Secondary Outcome: Summary of Changes in CD4% From Baseline to Week 48 (Cohort 2)
Description: The mean difference is calculated as CD4% at Week 48 minus CD4% at Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 48.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 48 timepoints.
Measure: Mean (95% Confidence Interval); unit: Percent of total lymphocytes
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 43
Percent of total lymphocytes |  | -0.4 [-1.7 to 0.9]

34. Secondary Outcome: Summary of Changes in CD4% From Baseline to Week 96 (Cohort 2)
Description: The mean difference is calculated as CD4% at Week 96 minus CD4% at the Day 0 with associated 95% Clopper-Pearson CI.
Time Frame: Measured at Day 0 and week 96.
Population: Cohort 2 participants who had non-missing values at both Day 0 and Week 96 timepoints.
Measure: Mean (95% Confidence Interval); unit: Percent of total lymphocytes
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 38
Percent of total lymphocytes |  | -0.5 [-2.5 to 1.5]

35. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events Assessed as Related to Study Drug (Cohort 2) Through End of Study
Description: Percentage and Clopper-Pearson 95% CI of participants with Grade 3 or higher AEs judged by the medical clinic as related to the study drug. AEs were graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017 (DAIDS) AE Grading table corrected version 2.1 (see References).
Time Frame: Measured from Day 0 through Week 96.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 45
Percentage of participants |  | 0 [0 to 7.9]

36. Secondary Outcome: Percentage of Participants With Serious Adverse Events Assessed as Related to Study Drug (Cohort 2) Through End of Study
Description: as for outcome 5
Time Frame: Measured from Day 0 through Week 96.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 45
Percentage of participants |  | 0 [0 to 7.9]

37. Secondary Outcome: Percentage of Participants With Permanent Discontinuation of Study Drug Due to Adverse Events Assessed as Related to Study Drug (Cohort 2) Through End of Study
Description: as for outcome 6
Time Frame: Measured from Day 0 through Week 96.
Population: Study Participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 45
Percentage of participants |  | 0 [0 to 7.9]

38. Secondary Outcome: Percentage of Participants With Grade 5 Adverse Events (Death) Regardless of Relationship to Study Drug (Cohort 2) Through End of Study
Description: Percentage and Clopper-Pearson 95% CI of participants with Grade 5 adverse events (death).
Time Frame: Measured from Day 0 through Week 96.
Population: Study participants who received at least one dose of study treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
Number analyzed (Participants) | 0 | 45
percentage of participants |  | 0 [0 to 7.9]

ADVERSE EVENTS:
Time Frame: From start of study treatment to study completion at Week 2 in Cohort 1 or at Week 96 in Cohort 2.
Description: AEs were summarized for participants who received at least one dose, and included abnormal laboratory events with specimen collection dates greater than first dose date and AEs that are not abnormal laboratory events and have onset dates equal to or greater than study drug's first dose date. AES were restricted to those with start dates less than or equal to the PCD. AE severity grading was based on the DAIDS AE Grading Table, Corrected Version 2.1. SAE were graded using DAIDS EAE Manual V2.0.
Groups:
- Cohort 2: DOR/3TC/TDF: Participants received DOR/3TC/TDF from Day 0 through Week 96. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF): DOR/3TC/TDF administered orally as a fixed-dose combination (as a tablet, 100 mg/300 mg/300 mg) once daily.
Arm/Group | Cohort 1: DOR | Cohort 2: DOR/3TC/TDF
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/45
Other Adverse Events (participants affected / at risk) | 4/9 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DOR (N=9) | Cohort 2: DOR/3TC/TDF (N=45)
COVID-19 (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DOR (N=9) | Cohort 2: DOR/3TC/TDF (N=45)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Flatulence (Gastrointestinal disorders) | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary gland mucocoele (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 0 | 3
Hordeolum (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 4
Pharyngitis (Infections and infestations) | 0 | 2
Pharyngitis bacterial (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Urethritis gonococcal (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Adverse event following immunisation (Injury, poisoning and procedural complications) | 0 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 21
Aspartate aminotransferase increased (Investigations) | 2 | 15
Blood albumin decreased (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 14
Blood bicarbonate decreased (Investigations) | 0 | 12
Blood bilirubin increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 7
Blood creatinine increased (Investigations) | 0 | 21
Blood glucose decreased (Investigations) | 0 | 6
Blood glucose increased (Investigations) | 1 | 8
Blood phosphorus decreased (Investigations) | 0 | 4
Blood phosphorus increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 9
Blood potassium increased (Investigations) | 0 | 2
Blood pressure increased (Investigations) | 0 | 8
Blood sodium decreased (Investigations) | 0 | 7
Blood triglycerides increased (Investigations) | 0 | 3
Carbon dioxide decreased (Investigations) | 0 | 11
Creatinine renal clearance decreased (Investigations) | 0 | 2
Glomerular filtration rate decreased (Investigations) | 0 | 25
Haemoglobin decreased (Investigations) | 0 | 7
Lipase increased (Investigations) | 0 | 8
Low density lipoprotein increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 3
Platelet count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone callus excessive (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Anosmia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 9
Lethargy (Nervous system disorders) | 0 | 1
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Tension (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 3
Glycosuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 6
Urethral discharge (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Bleeding anovulatory (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1
Penile swelling (Reproductive system and breast disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03332095/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03332095/SAP_002.pdf
  • Informed Consent Form (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03332095/ICF_000.pdf